CLINICAL TRIAL: NCT01834183
Title: A Phase II and Biomarker Study of Tivozanib With Gemcitabine Addition Upon Progression in Patients With Metastatic Refractory Renal Cell Carcinoma
Brief Title: Tivozanib + Gemcitabine in Metastatic RCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Aveo has withdrawn support for this trial.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Toni Choueiri, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-084
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — tivozanib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tivozanib/Gemcitabine (Experimental): Segment 1: Tivozanib, taken orally days 1-21 of each 28 day cycle. Segment 2: Tivozanib, taken orally days 1-21 of each 28 day cycle. Gemcitabine, taken intravenously, Days 1 and 8 of each 28 day cycle.
  Interventions: Drug: Tivozanib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Tivozanib
  Other Names: AV-951
Drug: Gemcitabine

SUMMARY:
This research study is a PHase II clinical trial, which tests the safety and effectiveness of an investigational combination of drugs to learn whether the combination of drugs works in treating a specific cancer. "Investigational" means that the combination of drugs is being studied. It also means that the FDA has not yet approved these drugs or combination of drugs for use in participants, including people with your type of cancer.

Tivozanib is an anti-angiogenesis medicine that fights cancer by cutting off a tumor's blood supply so that it does not get the blood and nutrients it needs to grow. This drug has been used in other research studies and information from those other research studies suggests that this drug may help to slow the growth of cancer cells.

Gemcitabine is a chemotherapy drug that is approved by the FDA for the treatment of pancreatic cancer and several other cancers. It is not approved for the treatment of renal cell carcinoma. Previous research suggests combining gemcitabine with tivozanib may have some effectiveness in treating metastatic renal cell carcinoma.

The purpose of this research study is to determine the effectiveness of tivozanib as a treatment for renal cell carcinoma. The purpose of this research study is to also determine if the combination of tivozanib and gemcitabine is effective in treating your type of cancer if your cancer becomes unresponsive or gets worse with tivozanib as treatment alone. The safety of the combination of tivozanib and gemcitabine will also wbe studied.

Another goal of this research study is to learn more about how tivozanib alone and the combination of tivozanib and gemcitabine may work to treat renal cell carcinoma. During the research study we will perform blood tests to measure the level of substances in the blood such as proteins (biomarkers) that may predict who will respond to treatment with tivozanib and gemcitabine.

DETAILED DESCRIPTION:
If you agree to participate in this study you will be asked to undergo some screening tests and procedures to confirm that you are eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in this study. If you have had some of these tests and procedures recently, they may or may not need to be repeated. The screening process will include the following: medical history, physical examination, measurement of vital signs, performance status assessment, electrocardiogram (EKG), echocardiogram (ECHO), CT or MRI, routine blood tests, urine sample, blood pregnancy test. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

This study is broken into two segments. In the first segment, you will receive tivozanib alone. Every 28 days in this study is called a study "cycle". You will come to clinic once every 28 days (once a month), on 'day 1' of each 28 day cycle.

Tivozanib is a pill that you take by mouth. You will take it once per day, in the morning, with a glass of water, with or without food. You will take tivozanib days 1-21 (the first three weeks) of each 28 day treatment cycle. You will be given a Study Drug Administration Diary to keep a brief record of the date and time when you take your dose of tivozanib. The study staff will explain to you how to complete your diary. This will be reviewed during yur visits by your doctor or a member of the study staff. This diary will be collected at your visit at the end of each cycle, and a new one will be given to you at the start of the next cycle. You will also have a pre-dose research blood draw (approximately 8 teaspoons of blood will be drawn) prior to your first dose of tivozanib, and after your first cycle of tivozanib. Your samples will not have personal information about you (such as your name and address) on them.

On Day 1 of every cycle you will have: a medical history, physical exam, measurement of your vital signs, performance status assessment, routine blood tests to monitor your health, urine sample. Every other cycle (prior to cycle 3, 5, 7 etc). you will have a CT or MRI scan, EKG, ECHO.

If your cancer gets worse while receiving tivozanib alone you may be eligible to participate in segment 2 of the study and receive tivozanib in combination with gemcitabine. You will come to the clinic on days 1 and 8 of each 28 day cycle.

Gemcitabine will be given through a vein (intravenously, or IV) over a period of 30 minutes at the study clinic. This is called an infusion. You will receive the gemcitabine on days 1 and 8 of each treatment cycle.

You will also have a pre-dose research blood draw (approximately 8 teaspoons of blood will be drawn) prior to your first cycle of tivozanib and gemcitabine in combination, after your first 28 days cycle of tivozanib and gemcitabine in combination, and if your cancer gets worse while receiving tivozanib and gemcitabine in combination. Your samples will not have personal information about you (such as your name and address) on them.

If your doctor determines it is safe for you to have a biopsy, you will undergo a fresh tumor biopsy at the following time points: Prior to receiving your first 28 day cycle of tivozanib and gemcitabine in combination; and after two 28 day cycles (roughly 2 months) of receiving tivozanib and gemcitabine in combination.

On Days 1 and 8 and at the end of study treatment you will undergo a medical history, physical examination, measurement of vital signs, performance status assessment, routine blood tests and a urine sample.

If an unexpected or unwanted event happens during the study, you may be asked to have some extra tests or measurements. Some of the tests or measurements done during the study may have to be repeated if the results are not usable or are abnormal. If additional visits are required during your participation in this study, your study doctor may perform the following procedures and evaluations: medical history, vital sign measurements, physical exam, ECG, performance status, blood and urine tests and/or a review of your study drug administration diary.

We would like to keep track of your medical condition indefinitely. If we do not hear from you, we would like to do this by calling no more than every three months to see how you are doing. Keeping in touch with you and checking your condition helps us look at the long-term effects of the research.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma that is metastatic
* Failed at least one prior VEGF-targeted therapy
* Prior immunotherapy and mTOR inhibitors are allowed
* Evidence of unidimensionally measurable disease based on RECIST 1.1 criteria, with at least 1 measurable lesion
* Willing to use adequate contraceptive measures while on study and for 30 days after the lst dose of study drug
* For Segment 2, must have evidence of progressive disease
* For Segment 2, amenable to start Gemcitabine chemotherapy within 6 weeks of progression on Tivozanib
* For Segment 2, willing to undergo pre/post therapy biopsy of a metastatic lesion if safe and amenable

Exclusion Criteria:

* Prior gemcitabine or tivozanib
* Anticipated need for major surgical procedure during the course of the study
* Pregnant or breastfeeding
* Known prior history of hypertensive crisis or hypertensive encephalopathy
* Primary central nervous system malignancies or leptomeningeal metastases
* Significant cardiac disease
* Subjects on warfarin
* Uncontrolled intercurrent illness
* Evidence of bleeding diathesis or known coagulopathy
* Serious, non-healing wound, ulcer or bone fracture
* Psychiatric illness/social situation that would limit compliance with study requirements
* Previous or concurrent malignancy requiring active systemic therapy, < 4 years
* Inability to swallow pills, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of tivozanib, major resection of the stomach or small bowel, or gastric bypass procedure
* Ongoing use of strong CYP3A4 inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate Activity and Toxicity of Tivozanib in mRCC Subjects | 2 years
  To evaluate the activity and toxicity of tivozanib in mRCC study participants who failed at least 1 prior VEGF-targeted therapy.

SECONDARY OUTCOMES:
Evaluate Activity and Toxicity of adding Gemcitabine in Subjects who Progress on Tivozanib | 2 years
  To evaluate the activity and toxicity upon adding gemcitabine in study participants who progress on tivozanib
Investigate Potential Biomarkers of Resistance to Tivozanib | 2 years
  To investigate potential biomarkers of resistance to tivozanib from metastatic RCC lesions and plasma at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Toni Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts